CLINICAL TRIAL: NCT06757686
Title: Evaluation of Maxillary Posterior Teeth Intrusion by Skeletally Anchored Mousetrap Appliance in Adult Patient With Anterior Open Bite
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MansouraU
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-08

CONDITIONS: Maxillary Molar Intrusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- maxillary molar intrusion (Experimental)
  Interventions: Device: Mousetrap appliance

INTERVENTIONS:
Device: Mousetrap appliance — two mini-implant will be inserted in the palate. then, the mousetrap appliance will be inserted on the mini-implant and activated with power chain.

SUMMARY:
Aim of the study: This clinical study aims to evaluate the dental, skeletal, and soft tissue effects of the Mousetrap appliance on the intrusion of maxillary posterior teeth in adult patients with anterior open bite.

Material and methods: An uncontrolled clinical trial will be conducted involving 20 participants aged 15 to 27 years with skeletal Class I, II, or mild Class III relationships and a measured AOB of 3-8 mm. Participants will receive mini-implants inserted in the anterior palate, with the Mousetrap appliance designed to promote molar intrusion while maintaining vertical dimension. Intraoral scans, radiographs, and clinical photographs will be recorded at baseline and post-intrusion.

DETAILED DESCRIPTION:
Aim of the study:

This clinical study will evaluate the dental, skeletal and soft tissue effects of skeletally anchored mousetrap appliance on the intrusion of maxillary posterior teeth in adult patient with anterior open bite.

Materials and methods:

Trial Design: This study will be uncontrolled clinical trial. Intervention All patients will start the treatment by mini-implants insertion in anterior palate. Application of topical and/or local anesthesia, mini-implants will be inserted in anterior palate, using a manual contra-angle driver. The implants are oriented perpendicularly to the palatal curvature. Intraoral scanning for maxillary arch will be recorded before and after intrusion for each patient; at T0 (before intrusion), T1 (after intrusion) appliance construction: the principle of the Mousetrap appliance. For molar intrusion, lever arms are connected to two mini-implants inserted in the anterior palate. A transpalatal arch is placed to avoid tipping of the molars during intrusion. Customized intrusion appliance including upper first molar with band and occlusal rest on posterior teeth. The appliance will be digitally designed. A modified transpalatal arch with a is fitted with sufficient clearance between the palatal mucosa to avoid impingement and irritation during and after successful molar intrusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 15 to 27 years.
* High angle patients with skeletal Class I, II or mild Class III.
* Patients with anterior open bite requiring maxillary posterior teeth intrusion as part of orthodontic treatment.
* Anterior open bite: range from 3-8 mm.
* Healthy adult patients.
* No previous orthodontic treatment.
* No evidence of either periodontal problems, gingival problems, or bruxism, at the beginning of orthodontic treatment.
* No medical problems interfering with orthodontic treatment.

Exclusion Criteria:

* Moderate to severe Class III skeletal relationship patients were excluded, as the molars intrusion would lead to increase the severity of Class III malocclusion.
* Patient with bad oral hygiene.
* Periodontal problems.

Ages: 15 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Amount of molar intrusion | 6 months
  The amount of molar intrusion performed, difference in the linear distance from the mesio-buccal cusp of maxillary first permanent molar to the palatal plane, between the pretreatment and post-intrusion cone-beam computed tomography records, will be measured

SECONDARY OUTCOMES:
external root resorption | 6 months
  To calculate the amount of external apical root resorption, each cusp tip and root apex will be precisely detected in all three planes (sagittal, coronal and axial), for all teeth included in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Mansoura university, Al Mansurah, Egypt